CLINICAL TRIAL: NCT06869174
Title: A Phase II Clinical Trial to Evaluate the Efficacy and Safety of Pucotenlimab in Combination with MRG002 in Treating HER2-positive Cancer of Unknown Primary
Brief Title: Pucotenlimab Combined with MRG002 for HER2-positive Cancer of Unknown Primary
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhiguo Luo, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Zhiguo Luo, MD, PhD, Proffessor, Fudan University
Organization: Fudan University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CUP 004
Record Dates: First submitted 2025-03-05; First posted 2025-03-11 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Cancer of Unknown Primary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Arm (Experimental)
  Interventions: Drug: Pucotenlimab combined with MRG002

INTERVENTIONS:
Drug: Pucotenlimab combined with MRG002 — Pucotenlimab 200mg iv d1, Q3W MRG002 2.2mg/kg d1, Q3W

SUMMARY:
This study is a single-arm, open-label, multicenter Phase II clinical trial designed to observe and evaluate the efficacy and safety of Pucotenlimab in combination with MRG002 in patients with HER2-positive (IHC 2+ or 3+) cancer of unknown primary.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form and comply with the protocol requirements.
2. Subjects must be ≥18 years of age on the day of signing the informed consent form, with no gender restrictions.
3. Expected survival of ≥3 months.
4. Subjects with histologically confirmed squamous cell carcinoma, adenocarcinoma, or undifferentiated carcinoma of unknown primary origin by pathology laboratory, and who also meet the criteria of HER2 immunohistochemistry (IHC) 2+ or 3+. Subjects must have received at least one line of systemic therapy, including but not limited to targeted therapy, immunotherapy, chemotherapy, etc.
5. Subjects must be able to provide a tumor specimen for pathological testing (paraffin block, paraffin-embedded sections, or fresh tissue sections are acceptable).
6. Radiological evidence of disease progression during or after the most recent treatment, as confirmed by the investigator; according to RECIST 1.1 criteria, at least one measurable lesion at baseline.
7. Adverse events (AEs) related to prior anti-tumor therapy must have resolved to ≤Grade 1 according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (NCI CTCAE v5.0), with the exception of alopecia, non-clinically significant or asymptomatic laboratory abnormalities.
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 within 7 days prior to dosing.
9. No severe cardiac dysfunction, with a left ventricular ejection fraction (LVEF) ≥50% within 28 days prior to dosing.
10. Adequate organ function.
11. Agree to contraception from the time of signing the informed consent form until 6 months after the last dose of the investigational drug. Women of childbearing potential must have a negative serum pregnancy test within 7 days before the first dose of the investigational drug.

Exclusion Criteria:

1. History of other primary malignancies.
2. Received prohibited treatments as per the protocol.
3. Untreated or unstable brain metastases, spinal metastases or compression, carcinomatous meningitis, or leptomeningeal metastases.
4. Presence of ascites, pleural effusion, pericardial effusion that cannot be controlled by drainage methods, or subjects who require drainage to control third-space effusions within 14 days before dosing.
5. Any severe or uncontrolled systemic disease, as judged by the investigator, including poorly controlled hypertension, uncontrolled diabetes, or signs of active bleeding.
6. History of uncontrolled cardiac disease, including heart failure greater than NYHA Class II, unstable angina, myocardial infarction within the past year, clinically significant supraventricular or ventricular arrhythmias requiring treatment, or prolonged QT syndrome.
7. Evidence of active infection, including hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) infection; uncontrolled active bacterial, viral, fungal, rickettsial, or parasitic infections, unless treated and resolved before administration of the investigational drug.
8. History of allergy to Pucotenlimab or any component of MRG002, or history of ≥Grade 3 allergic reaction to macromolecular protein preparations/monoclonal antibodies.
9. History of primary immunodeficiency or active autoimmune disease, current use of immunosuppressive agents, or systemic corticosteroid therapy (≥10 mg/day prednisone or equivalent), and continued use within 2 weeks before enrollment.
10. History of or concurrent interstitial pneumonia, severe chronic obstructive pulmonary disease, severe pulmonary insufficiency, symptomatic bronchospasm, etc.
11. Positive serum pregnancy test or breastfeeding women who do not agree to adequate contraception during the study and for 6 months after receiving the investigational drug.
12. Any other condition that, in the investigator's judgment, makes the subject unsuitable for participation in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-08 (Estimated); Primary Completion 2027-03-08 (Estimated); Study Completion 2028-08-08 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | Time from the date of recruiting to the first recorded complete remission (CR) or partial remission (PR), assessed up to 12 months.
  Defined as the percentage of participants in the analysis population who experienced a Complete Response or a Partial Response and was assessed using RECIST 1.1 based on investigator evaluation.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No